CLINICAL TRIAL: NCT06919055
Title: Biofeedback With Heart Sound Following Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Özcan (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Fatma Özcan, PhD Lecturer, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALLOSTAT0001
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Young Earthquake Survivors
Keywords: biofeedback, trauma, allostasis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Control group: 10 young 'healthy' earthquake survivors will not receive any auditory stimulation.
  1. Intervention group: 10 young 'healthy' earthquake survivors will be subjected to a closed circuit, real-time heart sound (PCG) (to create biofeedback).
  2. Intervention group: 10 young 'healthy' earthquake survivors will be given an auditory stimulus of their heart sound and average heart rate-MHR (or a metronome in heart rhythm) taken while calm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (Active Comparator): no stimulation during mental stress
  Interventions: Other: Control-no treatment
- PCG auditory stimulation group (Experimental): PCG auditory stimulation during mental stress
  Interventions: Other: PCG auditory stimulation
- metronome in heart rhythm stimulation group (Experimental): MHR (or a metronome in heart rhythm) stimulation during mental stress
  Interventions: Other: MHR stimulation

INTERVENTIONS:
Other: PCG auditory stimulation — PCG auditory stimulation during mental stress
  Arms: PCG auditory stimulation group
Other: MHR stimulation — MHR auditory stimulation during mental stress
  Arms: metronome in heart rhythm stimulation group
Other: Control-no treatment — no stimulation during mental stress
  Arms: control

SUMMARY:
The Project aims to assess the long-term risk of trauma-induced stress in young persons. Using non-invasive sound therapy to assess the effects on the vagal nerve via cardiovascular effects and neural activity will provide biofeedback in these individuals.

DETAILED DESCRIPTION:
Background: Some countries have suffered and will continue to suffer great destruction as a result of wars, epidemics, earthquakes, and other natural catastrophes. When individuals are exposed to specific psychological or physical traumas, they can develop stress-related disorders. This can lead to irreversible changes in the autonomic nervous system and cardiovascular disorders. When subjected to a new stress test, traumatized/previously exposed participants may show more pronounced behavioral changes, intolerance, and greater fatigue responses as compared to pre-trauma. To reduce trauma-associated responses from recurring again in the future, especially in young people, it is necessary to take preventive measures. Alternative solutions must be designed for counseling, medication, phytotherapy, etc. This study aims to examine how individuals cope with trauma-related situations using a biofeedback method, which could be developed to manage stress-related coping. The emotional and psychological states of earthquake victims will be assessed using a protocol based on biomedical (neuro-cardiac) signals and the sound of the person's own heart. This sound will be applied at a fixed frequency or in real-time with allostatic auditory stimulation. A resonance stabilizing the autonomic nervous system will thus provide biofeedback to the participants.

Methods: To examine the different states, biological signals will be measured and recorded, such as electrocardiography (ECG), phonocardiography (PCG), electrodermal activity, respiratory rhythm, and near-infrared spectroscopic imaging (fNIRS). Deep learning models will optimally process the collected data and evaluate the results.

Impact: The Project aims to assess the long-term risk of trauma-induced stress in young persons. Using non-invasive sound therapy to assess the effects on the vagal nerve via cardiovascular effects and neural activity will provide biofeedback in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* 30 earthquake survivor university students between 20 and 25 will participate in the experiment. Participants will be healthy, non-obese men (n=15) and women (n=15). In particular, all participants should have experienced the earthquake disaster in the local region. All participants must be free of any chronic or acute infection, neurological, psychiatric, and/or cardiovascular disease.

Exclusion Criteria:

* They must be non-smokers, have no alcohol or drug addiction, and not be under any medical treatment. Pregnant or breastfeeding women will not be included in the study.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 2 months
  In order to carry out this study, the following basic measurements (gender, age, height, weight, blood pressure, etc.) and relative measurements from the basic measurements will be extracted. In this context, earthquake victims' cardiological, emotional, and psychological states will be observed through biomedical signals.
  From electrocardiogram (ECG), HRV, LF, HF, LF/HF, SDNN, and RMSSD parameters will be assessed to evaluate the autonomic nervous system, especially the parasympathetic nervous system.
  The fNIRS device will measure changes in oxygenated and deoxygenated hemoglobin concentration in the cortical structure of the forebrain, as well as markers of cardiovascular and psychological risk.

SECONDARY OUTCOMES:
Others biopotentials | 2 months
  Our protocol will measure the electrodermal activity signal in microsiemens. The respiratory rythme is measured in milliVolt.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patron E, Calcagni A, Thayer JF, Scrimin S. The longitudinal negative impact of early stressful events on emotional and physical well-being: The buffering role of cardiac vagal development. Dev Psychobiol. 2021 Jul;63(5):1146-1155. doi: 10.1002/dev.22066. Epub 2020 Dec 11. PMID 33314062
- [Background] Parizek D, Visnovcova N, Hamza Sladicekova K, Veternik M, Jakus J, Jakusova J, Visnovcova Z, Ferencova N, Tonhajzerova I. Effect of Selected Music Soundtracks on Cardiac Vagal Control and Complexity Assessed by Heart Rate Variability. Physiol Res. 2023 Nov 28;72(5):587-596. doi: 10.33549/physiolres.935114. PMID 38015758
- [Background] Nakajima Y, Tanaka N, Mima T, Izumi SI. Stress Recovery Effects of High- and Low-Frequency Amplified Music on Heart Rate Variability. Behav Neurol. 2016;2016:5965894. doi: 10.1155/2016/5965894. Epub 2016 Aug 30. PMID 27660396
- [Background] Lee SW, Laurienti PJ, Burdette JH, Tegeler CL, Morgan AR, Simpson SL, Gerdes L, Tegeler CH. Functional Brain Network Changes Following Use of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology for Military-Related Traumatic Stress. J Neuroimaging. 2019 Jan;29(1):70-78. doi: 10.1111/jon.12571. Epub 2018 Oct 10. PMID 30302866
- [Background] Guannan, X., Xin, Z., Anchen, G., Siyang, H., Huijie, L., Jing, D., Qianqian, Z., & Jian, J. (2023). Phase-locked auditory pulse stimulation at home enhancing slow sleep waves: A pilot real-world study. medRxiv.
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Background] Fioranelli M, Bottaccioli AG, Bottaccioli F, Bianchi M, Rovesti M, Roccia MG. Stress and Inflammation in Coronary Artery Disease: A Review Psychoneuroendocrineimmunology-Based. Front Immunol. 2018 Sep 6;9:2031. doi: 10.3389/fimmu.2018.02031. eCollection 2018. PMID 30237802
- [Background] Adiasto K, Beckers DGJ, van Hooff MLM, Roelofs K, Geurts SAE. Music listening and stress recovery in healthy individuals: A systematic review with meta-analysis of experimental studies. PLoS One. 2022 Jun 17;17(6):e0270031. doi: 10.1371/journal.pone.0270031. eCollection 2022. PMID 35714120